CLINICAL TRIAL: NCT00693602
Title: Compassionate Use of Erwinase For Pediatric Patients With Acute Lymphoblastic Leukemia Or Non Hodgkins Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Jazz Pharmaceuticals (Industry); Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ERWASE
Record Dates: First submitted 2008-06-04; First posted 2008-06-09 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2011-12

CONDITIONS: Acute Lymphoblastic Leukemia; Non Hodgkins Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin | interventions — Asparaginase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Erwinase

INTERVENTIONS:
Drug: Erwinase — Chemotherapy

SUMMARY:
This is a compassionate use protocol for patients with acute lymphoblastic leukemia (ALL) who have developed hypersensitivity or intolerance to E. coli L-asparaginase and/or PEG-L-asparaginase.

DETAILED DESCRIPTION:
Primary Objective

To provide Erwinase to patients with acute lymphoblastic leukemia (ALL) or non-Hodgkins lymphoma who are intolerant or have developed hypersensitivity to E. coli asparaginase and/or PEG-asparaginase.

TREATMENT PLAN

Erwinia L-asparaginase administration will be given according to the protocol or non-protocol treatment plan under which the patient is currently being treated.

Erwinase will be discontinued in any patient experiencing an allergic reaction or any Grade 3 or higher adverse event believed to be attributable to this agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients on treatment for acute lymphoblastic leukemia or non-Hodgkins lymphoma receiving ALL-type therapy who have developed hypersensitivity or intolerance to E. coli L-asparaginase or PEG-L-asparaginase or both.
* Informed consent explained to and signed by parent/legal guardian, with emphasis that although approved for use in Europe and Canada, Erwinase is NOT approved by the United States Food and Drug Administration

Exclusion Criteria:

* Documented history of severe hypersensitivity or intolerance to Erwinase

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2006-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To provide Erwinase to patients with acute lymphoblastic leukemia (ALL) or non-Hodgkins lymphoma who are intolerant or have developed hypersensitivity to E. coli asparaginase and/or PEG-asparaginase | June 2009

CONTACTS AND LOCATIONS:
Overall Officials: Sima Jeha, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org